CLINICAL TRIAL: NCT03953794
Title: Inflammatory Bowel Disease Tracker (IBD Tracker)
Acronym: IBDTr
Status: Withdrawn | Type: Observational
Why Stopped: No accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Ashwin Ananthakrishnan, Assistant Professor of Medicine, Massachusetts General Hospital
Other Study IDs: 2017P002778
Record Dates: First submitted 2019-04-10; First posted 2019-05-17 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Optional blood, stool, and urine samples will be requested at various time points throughout the 12-month follow-up period. Optional biopsy samples can be collected at a standard-of-care endoscopic procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with inflammatory bowel disease: Patients who have...
  1. a diagnosis of ulcerative colitis or Crohn's disease as confirmed by a clinician
  2. experienced a flare within the past 24 months as determined by a clinician
  3. had quiescent disease for at least 3 months as determined by a clinician
  Interventions: Device: Fitbit Charge 3

INTERVENTIONS:
Device: Fitbit Charge 3 — Smart watch monitoring activity and movement, heart rate, sleep, and more

SUMMARY:
Inflammatory Bowel Diseases are incurable, life-long conditions that significantly impact a patient's quality of life. Crohn's Disease and ulcerative colitis are the most prevalent inflammatory bowel diseases in the United States; both are characterized by chronic, relapsing inflammation of the intestinal tract, which manifests as symptoms of diarrhea, fecal urgency, fecal incontinence, fever, fatigue, abdominal pain and cramping. These severely debilitating periods of illness or "flare" alternate with times of remission when patients have few or no symptoms, and feel healthy. Despite periodic respite, many patients with IBD experience severe stress and anxiety even when they are well, because of the likely occurrence of episodes of disease in their future. This is exacerbated by the unpredictable frequency and inconsistent duration of flares that may last as long as several weeks or months.

The goal for this study is to use non-invasive monitoring techniques to identify biomarkers that emerge, or change predictably, when a patient begins to relapse from remission to enter a period of disease - to find the earliest signs of an active flare. If the investigators identify a pattern of biomarkers that could alert a patient and their clinician to a flare as soon as it begins, it may be possible to intervene before symptoms present by changing medication and/or diet and lifestyle to lessen the severity of the disease flare. The biomarker fingerprint may also reveal new targets for therapeutics that could control IBD.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (IBD) is a chronic, incurable, life-long condition that significantly negatively impacts a patient's quality of life, and increases their risk of developing colorectal cancer. The causes of IBD are currently unknown, but are thought to be a combination of factors related to an individual's genetics, environment and immune system. A common characteristic of ulcerative colitis and Crohn's Disease, the most prevalent forms of IBDs in the United States, are chronic, relapsing inflammation of the intestinal tract. When patients are in remission they are healthy with no or few symptoms, and can lead normal and productive lives. However, these periods of health alternate with periods of illness (flares) with an unpredictable frequency, during which patients suffer from an array of symptoms including diarrhea, fecal urgency, fecal incontinence, fever, fatigue, abdominal pain and cramping. Inflammation in the colon and rectum often causes ulcers that bleed resulting in bloody stools; as inflammation continues, ulcers can get larger, and even join together increasing the volume of blood lost, leading to anemia in some cases. During episodes of active disease, patients experience a reduced appetite and unintended weight loss. Flares do not have a consistent duration, and can last from weeks to months. Symptoms can range from mild to severe, and can change over time.

According to the Centers for Disease Control and Prevention, there are currently an estimated 1-1.3 million people with IBD in the United States, and most of these patients are diagnosed with the disease before age 30. The burden of living with these lifelong conditions is obviously severe, however the financial burden should also be considered. In 2008, the total annual financial burden for direct treatments costs for patients with IBD in the United States was estimated to be $6.3 billion. Costs includes expenses such as physician services, prescription and over-the-counter drugs, hospitalization, and other direct medical expenses. Indirect costs (including lost earnings or productivity, and lost leisure time) were estimated to amount to an additional $5.5 billion.

Although the study is not targeted at finding a cure for IBD, the goal is to vastly improve the patient's quality of life by identifying biomarkers that emerge, or change predictably in a period leading up to the very beginning of a flare.

The investigators will identify biomarkers that predict an episode of disease is imminent. The investigators will target biomarkers that can be tracked non-invasively, by monitoring changes in the stool microbiome, metabolites in stool and urine, as well as physiological and lifestyle changes by asking patients to wear a wearable device (the Fitbit Charge 3). The investigators will collect blood samples regularly (blood draws are minimally invasive) to monitor additional biomarkers. By intensively monitoring patients in this way for a period of time that encompasses health (remission) and disease (flare), as well as the transition period in between, the investigators hope to amass enough data to tease out such a biomarker, or fingerprint of biomarkers, that benchmark the earliest stages of a flare. The investigators will conduct this study in collaboration with researchers at the Center for Microbiome Informatics and Therapeutics at Massachusetts Institute of Technology.

The ability to non-invasively track biomarkers, to monitor a patient for such an early disease fingerprint, may give that patient the power to manage their lives and their disease with greater precision than they can today. In particular, if that early disease fingerprint appears at a time when the patient still feels well, it is possible they could intervene to block progression of the flare by changing medications, and/or making lifestyle changes thus minimizing the impact of the flare, and the symptoms they experience.

Furthermore, pinpointing the molecular changes that occur systemically, throughout the patients during this transition period, from health (remission) to disease (flare) will give researchers the knowledge and tools with which to begin to develop therapies that can block progression of the disease state, preventing the flare, and perhaps "reset" the body to a state of health. Therapies, like these would greatly relieve the burdens of disease and financial costs for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to provide written informed consent prior to screening and willing to comply with the requirements of the study protocol
* Have had a diagnosis of ulcerative colitis or Crohn's Disease confirmed by a clinician
* Have had quiescent disease for the past 3 months or longer as determined by clinician
* Have had most recent episode of disease within past 24 months as determined by clinician
* Have had stable IBD medication (other than antibiotics) regimen for the past 3 months or longer
* Able to speak and read English sufficiently
* Be able and comfortable using new technology: the app and the smartwatch for 12 months

Exclusion Criteria:

* If female, is pregnant or is breast feeding, or intends to become pregnant within the 12 month study period
* Unable to provide informed consent or unwilling to participate
* Use of oral or intravenous antibiotics within 4 weeks prior to screening
* Current use of glucocorticoid steroid, or nonsteroidal anti-inflammatory drugs (NSAIDs) within the last 3 months
* Evidence of untreated infection e.g. Clostridium difficile
* Confirmed diagnosis of extraintestinal manifestations (EIMs) of disease including those that occur concurrent with colitis (episcleritis, scleritis, uveitis, peripheral arthropathies of small and large joints, dermatologic conditions such as erythema nodosum and pyoderma gangrenosum), and those that occur independent of colitis (sacroilitis, ankylosing spondylitis, or primary sclerosing cholangitis)
* Confirmed diagnosis of other serious disease unrelated to ulcerative colitis or Crohn's Disease
* Current smoker
* Unable to speak or read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with established inflammatory bowel disease who have had quiescent disease for at least 3 months but have experienced a flare within the last 24 months
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Simple Clinical Colitis Activity Index | 1 week
  Patient-reported measure for ulcerative colitis referring to disease symptoms occurring over the last week. The point value from each answer is added up for a total score.
  1. Over the past week, what is your average number of bowel movements during the day (not including night)? (0) 0-3 (1) 4-6 (2) 7-9 (3) >9
  2. Over the past week, what is your average number of bowel movements at night? (0) 0 (1) 1-3 (2) >3
  3. Over the past week, what has been your urgency of defecation? (0) No rush (1) Hurry (2) Immediately (3) Incontinence
  4. Over the past week, what has been the amount and frequency of blood in your stool? (0) None (1) Small traces (2) Occasionally obviously bloody (3) Usually obviously bloody
  5. General well being (0) Very well (1) Slightly below par (2) Poor (3) Very poor (4) Terrible
  6. During the past week, have you had any of the following? (1 pt/answer) (1) Pyoderma gangrenosum (1) Erythema nodosum (1) Uveitis (1) Arthritis (0) None
Harvey-Bradshaw Index | 1 week
  Patient-reported measure for Crohn's disease referring to disease symptoms occurring over the last week. The point value from each answer is added up for a total score.
  1. General well being (0) Very well (1) Slightly below par (2) Poor (3) Very poor (4) Terrible
  2. In the past week, have you experienced any abdominal pain? (0) None (1) Mild (2) Moderate (3) Severe
  3. How many liquid stools do you pass per day? (1 point per liquid stool)
  4. Do you have an abdominal mass? (0) None (1) Dubious (2) Definite (3) Definite and tender
  5. During the past week, have you had any of the following? (1 point per answer) (1) Pyoderma gangrenosum (oozing ulcers, usually on the leg) (1) Erythema nodosum (red, swollen bumps, on the skin (1) Uveitis (red, painful eyes) (1) Aphthous ulcers (mouth ulcers) (1) Arthritis (joint pain) (1) Anal fissue (1) New fistula (1) Perianal abscess (0) None of the above
Stress and Wellbeing | Current moment in time
  Patient-reported measure of current stress level measured on a scale of 1 (1 = no stress) to 5 (5 = highest stress possible)
24-hour dietary recall survey | 24 hours
  Patient-reported measure of diet over the last 24 hours. The survey can be found here: https://asa24.nci.nih.gov/demo/
Blood biomarkers - metabolite content | 12 months
  Metabolite content will be determined by monitoring patients via regular blood draws over the 12-month study period. By analyzing metabolite content in periods of health (remission), disease (flare), and the transition period in between, investigators hope to identify unique biomarkers that indicate the earliest stages of a flare. The investigators do not know each specific metabolite that will be measured. The objective of this outcome is to identify any and all possible biomarkers and metabolites that may be present in these samples.
Blood biomarkers - cytokine profile | 12 months
  Cytokine profile will be determined by monitoring patients via regular blood draws over the 12-month study period. By analyzing cytokine profile in periods of health (remission), disease (flare), and the transition period in between, investigators hope to identify unique biomarkers that indicate the earliest stages of a flare. The investigators do not know each specific biomarker and cytokine that will be measured. The objective of this outcome is to identify any and all cytokines that may be present in these samples.
Blood biomarkers - T-cell receptor sequence profile | 12 months
  T-cell receptor sequence profiles will be determined by monitoring patients via regular blood draws over the 12-month study period. By analyzing T-cell receptor sequence profiles in periods of health (remission), disease (flare), and the transition period in between, investigators hope to identify unique biomarkers that indicate the earliest stages of a flare.
Stool biomarkers - microbial DNA content in microbiome | 12 months
  Patients will submit weekly stool samples for analysis and monitoring. The investigators will analyze the gut microbiome composition by characterizing the microbial DNA content and tracking changes throughout the 12-month study period. The investigators do not know each microbe that will be assessed. The objective of this outcome is to identify any and all microbes that may be present in these samples.
Stool biomarkers - overall microbiome content | 12 months
  The investigators will analyze the bacterial, fungal, and viral constituents at enrollment and and track changes throughout the 12-month study period to identify biomarkers of importance. These will be assessed with stool wipe samples, glycerol-preserved stool, and fresh and ethanol-preserved stool samples. Stool samples will either collected by patients at home or collected in-clinic and flash frozen.
Stool biomarkers - degree of intestinal inflammation via Fecal Calprotectin | 12 months
  The investigators will measure the degree of intestinal inflammation by quantifying Fecal Calprotectin (a biomarker) levels in patients' weekly stool samples and tracking changes throughout the 12-month study period. This will be measured using stool wipe samples and fresh stool samples.
Urine biomarkers - metabolite content | 12 months
  The investigators will use urine samples collected throughout the study to analyze each subject's urine metabolite content and track changes throughout the 12-month study period in an attempt to identify biomarkers potentially indicative of a flare. The investigators do not know each specific metabolite that will be measured. The objective of this outcome is to identify any and all possible biomarkers and metabolites that may be present in these samples.

SECONDARY OUTCOMES:
Biospecimen association - microbiome timeseries and blood and stool metabolites | 12 months
  Investigators will measure any existing correlations between the microbiome timeseries and the identified blood and stool metabolites over the 12-month study period to determine if there are any associations between the two variables.
Biospecimen association - microbiome composition and fecal calprotectin levels | 12 months
  Investigators will measure any existing correlations between the microbiome composition and fecal calprotectin levels identified in the primary outcomes over the 12-month study period to determine if there are any associations between the two variables.
Biospecimen association - blood and stool metabolites and microbiome composition | 12 months
  Investigators will measure any existing correlations between the identified blood and stool metabolites and the microbiome composition over the 12-month study period to determine if there are any associations between the two variables.
Biospecimen association - stool metabolites and blood metabolites | 12 months
  Investigators will measure any existing correlations between the identified blood metabolites and the identified stool metabolites and the microbiome composition over the 12-month study period to determine if there are any associations between the two variables.

IPD SHARING:
Plan to Share IPD: Undecided